CLINICAL TRIAL: NCT05342701
Title: The CHAMP Afterschool Program: Promoting Physical Activity & Health in Children
Brief Title: The CHAMP ASP: Promoting Physical Activity & Health in Children
Acronym: CHAMP-ASP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Leah Robinson, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00208311; R01NR018830 (NIH)
Record Dates: First submitted 2022-03-16; First posted 2022-04-25 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHAMP-ASP (Experimental): CHAMP, is a mastery climate motor skills intervention, that provides children the opportunity to establish behaviors that reinforce decision-making while participating in a motor activity tasks. Children will participate in CHAMP for 35 minutes/day 3-4 days per week for 19 weeks.
  Each 35-min session consists of three parts:
  1. 3-5 min of motor skill introductory activity that includes a group motor activity, the teaching of the lesson that includes a demonstration and understanding of developmentally appropriate learning clues;
  2. 25 min of motor skill instruction and practice (i.e., 'active motor engagement'), participants will be encouraged to move through 3-4 motor activity stations that align with the TARGET structure; and
  3. 3 -5 min motor skill closure activity that involves a review of the lesson and critical elements.
  Interventions: Behavioral: Motor Skills Intervention
- Control - Standard of Practice (No Intervention): The Control (standard of practice) condition will be the school typical ASP and will be implemented according to the existing procedures.

INTERVENTIONS:
Behavioral: Motor Skills Intervention — The behavioral motor skill intervention (CHAMP) is an intervention strategy that uniquely address differences in children's development. CHAMP does not equate to a "one size fits all" approach. Children will be in an environment that promotes opportunities for them to development improvement in motor skills based on their specific individual needs and choices. The CHAMP intervention promotes a mastery climate that allows each individual child to be successful and learn while promoting intrinsic motivation and autonomy. CHAMP consists of 35 minutes/day X 3-4 days/week for 19 weeks (dose of 1995 - 2240 minutes). Each session will consist of three parts: (a) 3-5 min of motor skill introductory activity, (b) 25 min of motor skill instruction and practice, and (c) 3-5 min motor skill closure activity.
  Arms: CHAMP-ASP

SUMMARY:
Currently, 10 million children participate in afterschool programs (ASPs) each day, and ASPs provide a great opportunity to enhance children's health outside of the regular school environment, particularly given the decline in physical education. This proposed, randomized cluster, controlled trial will examine the immediate (pre- to post-test) and sustained (1-year post-intervention follow-up) effects of CHAMP-ASP on physical activity (primary outcome), motor performance, perceived motor competence, health-related physical fitness, and weight status. CHAMP-ASP will be implemented by ASP staff and will be conducted in ASPs located in Ypsilanti/Ann Arbor, Michigan. Children (N = 264; CHAMP-ASP=132 and control=132) K-2 graders (typically ages 5-8 years) will participate 35 minutes/day X 3-4 days/week for 19 weeks (dose of 1995 - 2240 minutes). The aims are to: a) examine the immediate and sustained effects of CHAMP-ASP on physical activity, motor performance, and perceived motor competence relative to the control ASP, b) examine the immediate and sustained effects of CHAMP-ASP on secondary health outcomes - health-related physical fitness (cardiorespiratory fitness, muscular strength), and weight status compared to children in schools randomized to control ASP, and c) determine if perceived motor competence mediates the effect of CHAMP-ASP on moderate-to-vigorous physical activity.

DETAILED DESCRIPTION:
Promoting health-enhancing and sustainable physical activity levels across childhood and adolescence contributes to adult health. The Children's Health Activity Motor Program (CHAMP) is an evidence-based intervention that demonstrates impactful results on motor performance, perceived motor competence, and physical activity in physical education and movement-based settings. Currently, 10 million children participate in afterschool programs (ASPs) each day, and ASPs provide a great opportunity to enhance children's health outside of the regular school environment, particularly given the decline in physical education. This proposed, randomized cluster, controlled trial will examine the immediate (pre- to post-test) and sustained (1-year post-intervention follow-up) effects of CHAMP-ASP on physical activity (primary outcome), motor performance, perceived motor competence, health-related physical fitness, and weight status. CHAMP-ASP will be implemented by ASP staff and will be conducted in ASPs located in Ypsilanti/Ann Arbor, Michigan. Children (N = 264; CHAMP-ASP=132 and control=132) K-2 graders (typically ages 5-8 years) will participate 35 minutes/day X 3-4 days/week for 19 weeks (dose of 1995 - 2240 minutes). The aims are to: a) examine the immediate and sustained effects of CHAMP-ASP on physical activity, motor performance, and perceived motor competence relative to the control ASP, b) examine the immediate and sustained effects of CHAMP-ASP on secondary health outcomes - health-related physical fitness (cardiorespiratory fitness, muscular strength), and weight status compared to children in schools randomized to control ASP, and c) determine if perceived motor competence mediates the effect of CHAMP-ASP on moderate-to-vigorous physical activity. The long-term goal is to provide a sustainable, ecologically-relevant, and evidence-based program during the early elementary years that is health-enhancing and increases physical activity in school-age children. Findings could significantly influence future physical activity interventions and support a sustainable, ecologically-relevant (delivered by ASP staff) evidence-based program (i.e., CHAMP) that contributes to long-term health-enhancing physical activity and health in children.

ELIGIBILITY:
Inclusion Criteria:

-Participants must be attending an ASP in the Ann-Arbor/Ypsilanti and Lansing/East Lansing area

Exclusion Criteria:

* Participants diagnosed with syndromes or diseases that affect PA participation
* Participants diagnosed with any major illness, developmental, and/or physical disability that limited their ability to participate in movement and physical activity programs.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 264 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Motor Competence - process measures | baseline, post-intervention (i.e., 24 weeks post baseline), and 1 year post-intervention follow-up
  Process scores will be assessed with the Test of Gross Motor Development (TGMD, 3rd edition); scores from the two subscales (locomotor and ball skills) will be reported as raw scores for each skills and an overall score (total MC score). The project will assess changes overtime for this measure
Changes in Motor Competence - product measures | baseline, post-intervention (i.e., 24 weeks post baseline), and 1 year post-intervention follow-up
  Product scores will use throwing speed, kicking speed, jump distance, running speed, and hopping speed. Product score will vary for each participant (i.e., kick, run, hopping, and throw velocity along with jumping distance - faster scores and greater distance are indicators of better MC).
Changes in Physical Activity | baseline, post-intervention (i.e., 24 weeks post baseline), and 1 year post-intervention follow-up
  Actigraph GTX3+ tri-axial accelerometer will be used to measure the frequency, intensity, and duration of PA among children during the ASP and in free-living settings. Participants will be asked to wear the same accelerometer for 7 full days (5 week and 2 weekend days). Data will be set to collect data in raw mode (30 Hz), and will be processed using ActiLife software or other, more advanced techniques, such as machine learning approaches.
Changes in Health-related fitness - Cardiorespiratory endurance | baseline, post-intervention (i.e., 24 weeks post baseline), and 1 year post-intervention follow-up
  Cardiorespiratory endurance will be assessed with a 6-min walk test. For the 6-min walk test, the children walk as fast as possible around two cones for 6 minutes.
Changes in Health-related fitness - Muscular Strength | baseline, post-intervention (i.e., 24 weeks post baseline), and 1 year post-intervention follow-up
  Muscular strength will be assessed with test of handgrip strength. Upper body strength will be assessed using a hand grip strength with a dynamometer, which has been deemed reliable and valid in 6-12-year-olds [62]. Grip will be appropriately adjusted for size, and two trials on the right and left sides (elbow extended) will be assessed (muscular strength). The sum of maximum score (kg) of two trials for each hand will be used in analyses.
Changes in Health-related fitness - Body Composition | baseline, post-intervention (i.e., 24 weeks post baseline), and 1 year post-intervention follow-up
  Body composition (i.e., body fat) will be assessed with bioelectrical impedance. Body fat percentage will be the average of two measurements assessed (to the nearest 0.1%, respectively) with a bioelectric impedance analysis scale (Tanita). The assessment will be completed in a designated, private area

SECONDARY OUTCOMES:
Demographics | Baseline
  Date of birth, sex, race/ethnicity, and grade will be collected through self-report through the IRB consenting process by the parent/guardian.
Changes in Perceived Motor Competence (Global) | baseline, post-intervention (i.e., 24 weeks post baseline), and 1 year post-intervention follow-up
  Will be assessed with the Harter and Pike Pictorial Scale of PMC and Social Acceptance (PSPCSA). The PSPCSA will be used to measure the child's global perceived physical competence. The PSPCSA physical competence subscale consists of six items that are presented in pictures and each child will select a picture that is more like them. The six items included are swinging, climbing, tying shoe laces, skipping, running, and hopping. For the assessment, children will (1) select the picture that is most like him or herself. One picture depicts a child who is competent and the other shows a child who is not skilled; (2) focus on the designated pictures and indicate whether he or she is just a "little bit" or "a lot" like that child. Separate pictures for girls and boys will be used in accordance with the manual procedures. The range of scores for each item on the subscale is 1 (low competence) to 4 (high competence).
Changes in Digital Scale of Perceived Motor Competence (DSPMC) | baseline, post-intervention (i.e., 24 weeks post baseline), and 1 year post-intervention follow-up
  Will be assessed with the Digital Scale of Perceived Motor Competence (DSPMC) The DSPMC is a video-based assessment that allows the child to see the entire motor skill in action (video) rather than a static picture. The scale is the identical layout and item structure to the PSPCSA but align with the 12 fundamental motor skills of the TGMD For the assessment, children will (1) select the video that is most like him or herself. One video depicts a child who is competent and the other shows a child who is not skilled; (2) focus on the designated videos and indicate whether he or she is just a "little bit" or "a lot" like that child. The range of scores for each item on the subscale is 1 (low competence) to 4 (high competence).
CHAMP ASP Acceptability Questionnaire | post-intervention (i.e., 24 weeks post baseline)
  Children will complete an acceptability survey to provide information on how they like participating in the CHAMP-ASP program. The CHAMP-ASP Acceptability Questionnaire consists of 6 questions about the program's features such as children's autonomy to determine for how long they want to be doing the selected activity and how the ASP staff provided them feedback. For each question the child will answer with yes or no.
Family Questionnaire | baseline
  Parents will be asked to complete a family questionnaire to provide some descriptive information about their child and family. Questions are regarding the family structure, socio-economic status, physical activity habits, sleeping habits, and screen time habits. The questionnaire has closed ended questions that will be quantified for data analyses.
Changes Social-emotional measure | baseline, post-intervention (i.e., 24 weeks post baseline), and 1 year post-intervention follow-up
  Parents will be asked to complete the Strength and Difficulties Questionnaire (SDQ) which is a relatively short instrument developed to screen for emotional and behavioural problems in children aged 3-16 years [59]. The SDQ is a 25-item questionnaire with three response categories from zero to two (not true, somewhat true, and certainly true). The questionnaire has five subscales of five items each: emotional problems, conduct problems, hyperactivity/inattention problems, peer problems, and prosocial behaviour.
Changes in Body Mass Index | baseline, post-intervention (i.e., 24 weeks post baseline), and 1 year post-intervention follow-up
  Will be used to calculate body mass index (BMI) with height and weight will be assessed with the participant barefoot and in light clothing. Standing height will be measured to the nearest 0.1 cm using a portable stadiometer and the average of two measurements to the nearest 0.1 cm (Shorr Productions, Olney, MD). Weight will be the average of two measurements assessed (to the nearest 0.1 kg and 0.1%, respectively) with a weight scale. BMI will be calculated, and, using age and sex and the CDC growth charts,95 transformed into BMI z-score for analyses. The assessment will be completed in a designated, private area

CONTACTS AND LOCATIONS:
Overall Officials: Leah E Robinson, PhD, Principal Investigator — University of Michigan
Locations (1):
- Leah Elizabeth Robinson, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lohman TG, Ring K, Pfeiffer K, Camhi S, Arredondo E, Pratt C, Pate R, Webber LS. Relationships among fitness, body composition, and physical activity. Med Sci Sports Exerc. 2008 Jun;40(6):1163-70. doi: 10.1249/MSS.0b013e318165c86b. PMID 18460987
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] Robinson LE, Palmer KK, Bub KL. Effect of the Children's Health Activity Motor Program on Motor Skills and Self-Regulation in Head Start Preschoolers: An Efficacy Trial. Front Public Health. 2016 Sep 8;4:173. doi: 10.3389/fpubh.2016.00173. eCollection 2016. PMID 27660751
- [Background] Robinson LE, Veldman SLC, Palmer KK, Okely AD. A Ball Skills Intervention in Preschoolers: The CHAMP Randomized Controlled Trial. Med Sci Sports Exerc. 2017 Nov;49(11):2234-2239. doi: 10.1249/MSS.0000000000001339. PMID 29045324
- [Background] Robinson LE, Stodden DF, Barnett LM, Lopes VP, Logan SW, Rodrigues LP, D'Hondt E. Motor Competence and its Effect on Positive Developmental Trajectories of Health. Sports Med. 2015 Sep;45(9):1273-1284. doi: 10.1007/s40279-015-0351-6. PMID 26201678
- [Background] Beets MW, Beighle A, Erwin HE, Huberty JL. After-school program impact on physical activity and fitness: a meta-analysis. Am J Prev Med. 2009 Jun;36(6):527-37. doi: 10.1016/j.amepre.2009.01.033. Epub 2009 Apr 11. PMID 19362799
- [Background] Lima RA, Pfeiffer K, Larsen LR, Bugge A, Moller NC, Anderson LB, Stodden DF. Physical Activity and Motor Competence Present a Positive Reciprocal Longitudinal Relationship Across Childhood and Early Adolescence. J Phys Act Health. 2017 Jun;14(6):440-447. doi: 10.1123/jpah.2016-0473. Epub 2017 Feb 7. PMID 28169569
- [Derived] Robinson LE, Palmer KK, Santiago-Rodriguez ME, Myers ND, Wang L, Pfeiffer KA. Protocol for a multicenter-cluster randomized clinical trial of a motor skills intervention to promote physical activity and health in children: the CHAMP afterschool program study. BMC Public Health. 2022 Aug 13;22(1):1544. doi: 10.1186/s12889-022-13849-8. PMID 35964114

DOCUMENTS (1):
  • Informed Consent Form (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT05342701/ICF_000.pdf